CLINICAL TRIAL: NCT06459648
Title: Prediction Study or Response to Treatment With Anti-CGRP Monoclonal Antibodies in Migraine
Brief Title: Study for Prevent Chronification Migraine Through Prediction of Response to Treatment With Anti-CGRP Antibodies
Acronym: PREDI-CGRP
Status: Recruiting | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Other Study IDs: PI 23- 3054
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Migraine
Keywords: Migraine; headache; antibodies; antibody; monoclonal antibody; anti-cgrp; anti cgrp; cgrp; prediction; treatmen; migraine treatment; treatment with anti-CGRP monoclonal antibodies; anti-cgrp antibodies; anti-cgrp antibody; anti-cgrp monoclonal antibodies; migraine and antibodies; migraine and cgrp
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — The samples collected from the patients in the study are blood and neuroimaging samples, specifically, brain MRIs without contrast. Thanks to the blood samples, serum, plasma as well as peripheral blood mononuclear cells (PBMCs) will be analyzed. This analysis will allow measurement of CGRP levels in blood, genome sequencing to obtain the genotype of each participant and estimate their polygenic risk of disease, methylome sequencing to obtain the methylation profile of the CpG islands described in human chips and finally data of transcriptomics, specifically miRNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with migraine under treatment with monoclonal antibodies against CGRP: Patients with diagnosis of episodic or chronic migraine who, under the criteria of their neurologist and according to the clinical practice guidelines and standard of care, receive treatment with monoclonal antibodies against CGRP (Galcanezumab, Fremanezumab, Eptinezumab) or else its receptor (Erenumab) will be included.
  Interventions: Other: Headache record; Other: Scales; Drug: Monoclonal antibody anti-CGRP

INTERVENTIONS:
Other: Headache record — The patient will keep a record of the presence/absence of headache, average intensity, and need for acute medication.
Other: Scales — Each patient performs different scales that measure the impact of the migraine on their daily life as well as the disability it may be causing. In turn, each patient performs different scales that measure associated comorbidities such as depression, anxiety or insomnia.
Drug: Monoclonal antibody anti-CGRP — Erenumab, Galcenazumeb, Fremanezumab, Eptinezumab

SUMMARY:
Being able to predict each patients response to a specific treatment can mean a significant improvement in socioeconomic costs, but above all in their quality of life. With the present study, the investigators aim to analyze in a combined way different clinical, biological and neuroimaging variables, which allow the clinical staff to anticipate the response to treatment with anti-CGRP monoclonal antibodies in patients with migraine.

DETAILED DESCRIPTION:
The study consists of an initial visit coinciding with the start of treatment, a subsequent visit after 6 months of treatment and finally another after 12 months, coinciding with the end of treatment. In case of worsening after suspension, a clinical visit will be carried out at the time of worsening to evaluate the reintroduction of the drug and in case of reintroduction, a visit will be carried out after 3 months. If patients do not worsen, a visit will be made 6 months after completing treatment.

At each visit, demographic and clinical variables will be collected. In addition, 3 blood tests will be performed corresponding to the beginning of treatment, after 6 months and a month and a half from the last infiltration. Likewise, a brain MRI will be obtained prior to the start of treatment. These blood samples and neuroimaging data will be processed for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years.
* Caucasian ethnicity.
* Patients diagnosed with migraine with and without high-frequency episodic aura (more than 8 days of migraine per month) or chronic by a neurologist expert in headaches and according to the criteria proposed in the International Classification of Headache Diseases, 3rd edition (ICHD- 3).
* Have at least one year of history of migraine.
* Patients must maintain stable preventive treatment in the previous month and not have received botulinum toxin in the month prior to starting the monoclonal antibody.
* Patients able to describe their clinical situation and the characteristics of their headache.
* Grant your informed consent.

Exclusion Criteria:

* Patients who present with another type of non-migraine headache, with the exception of headache due to excessive use of analgesic medication.
* Neurological focus in the examination.
* Pregnancy or breastfeeding period.
* Patients with cognitive deficiency or pathology that may prevent or hinder the correct completion of the study.
* Patients who require changes in preventive treatment during the first 6 months after starting treatment with monoclonal antibodies.
* Patients who present any significant adverse effect that requires withdrawal or change of anti-CGRP drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 65 years with a diagnosis of episodic or chronic migraine who, at the discretion of their neurologist and according to clinical practice guidelines and standard of care, receive treatment with monoclonal antibodies against CGRP (Galcanezumab, Fremanezumab, Eptinezumab) or its receptor (Erenumab) be included. These patients will come from 7 Headache Units in Spain belonging to the following hospitals:
  * La Princesa University Hospital
  * Vall d'Hebron University Hospital
  * Marqués de Valdecilla University Hospital
  * Valladolid University Clinical Hospital
  * Donostia University Hospital
  * Lozano Blesa University Clinical Hospital
  * La Fe Polytechnic University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of positive initial response to monoclonal antibodies | From the beginning of treatment, which is the initial visit, to 18 months of follow-up
  Establish clinical, demographic, transcriptomic, genetic, molecular and/or radiological characteristics that allow predicting a positive initial response to monoclonal antibodies (biomarkers of therapeutic response).

SECONDARY OUTCOMES:
Sustained response factors | From the beginning of treatment, which is the initial visit, to 18 months of follow-up
  To analyze sustained response factors at the sociodemographic, clinical, transcriptomic, genetic, molecular and/or radiological level after the suspension of anti-CGRP drugs.
Sustained response after discontinuation of the anti-CGRP antibody | From the beginning of treatment, which is the initial visit, to 18 months of follow-up
  To quantify the proportion of patients who present a sustained response after discontinuation of the anti-CGRP antibody.
Non-maintained pharmacological response relation with biomarkers | From the beginning of treatment, which is the initial visit, to 18 months of follow-up
  To characterize whether the non-maintained pharmacological response is related to the variables previously characterized as predictors of chronicity.
Time until relapse after discontinuation of the anti-CGRP antibody | From the beginning of treatment, which is the initial visit, to 18 months of follow-up
  To determine the time until relapse after discontinuation of the anti-CGRP monoclonal antibody in those patients who, having presented a positive initial response, discontinue it.
Biomarkers of patients with high-frequency episodic migraine and chronic migraine | From the beginning of treatment, which is the initial visit, to 18 months of follow-up
  To validate possible transcriptomic, genetic, molecular and/or radiological characteristics that allow differentiation between patients with high-frequency episodic migraine and chronic migraine in a national multicenter cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Beatriz Gago Veiga, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (7):
- Spain (7):
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Universitari Vall d'Hebron Research Institute, Barcelona, Catalonia
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Universitario Politécnico La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon reasonable request to the principal investigator.